CLINICAL TRIAL: NCT06029439
Title: Long-term Study to Assess the Safety and Effectiveness of NMRA-335140 in Participants With Major Depressive Disorder
Brief Title: Study to Assess the Safety and Effectiveness of NMRA-335140-501
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neumora Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMRA-335140-501; KOASTAL-LT (Other: Neumora Therapeutics)
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; NMRA-335140; Long-term; Safety; Efficacy; Navacaprant; NMRA335140; NMRA 335140
MeSH Terms: conditions — Depressive Disorder, Major | interventions — BTRX-335140

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NMRA-335140 80 milligrams (mg) once daily (QD) (Experimental): Participants will receive a NMRA-335140 tablet at a dose of 80 mg once daily (QD) during a 52-week treatment period.
  Interventions: Drug: NMRA-335140

INTERVENTIONS:
Drug: NMRA-335140 — Participants will receive NMRA-335140 at a dose of 80 mg once daily (QD), orally during a 52-week treatment period.
  Other Names: BTRX-335140; CYM-53093; Navacaprant

SUMMARY:
This is a 52-week open-label extension (OLE) study that will evaluate the safety, tolerability, and effectiveness of NMRA-335140 in participants with major depressive disorder (MDD). Participants who completed a parent study investigating the efficacy and safety of NMRA-335140 as a treatment for MDD (ie, NMRA-335140-301, NMRA-335140-302, or NMRA-335140-303), and complete the 6 weeks double-blind treatment, provide informed consent, and meet eligibility criteria, may enter this extension study.

ELIGIBILITY:
Key Inclusion Criteria:

Rollover participants are eligible for the study if the following inclusion criteria are met:

* Completed a previous NMRA-335140 Phase 3 MDD study (example: NMRA-335140-301, NMRA-335140-302, or NMRA-335140-303) according to the completion definition in the parent study protocol.
* Signed an informed consent form (ICF) for this study.
* Willing to comply with the contraception requirements described in the inclusion criteria of the parent study protocol.
* Willing to comply with the concomitant medication/therapy restrictions described in the exclusion criteria of the parent study protocol.

Key Exclusion Criteria:

Rollover participants are excluded from the study if any of the following exclusion criteria are met:

* Diagnosed with another Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) disorder that would have been exclusionary in the parent study (eg, personality disorder, bipolar 1 or 2, schizophrenia, any other psychotic disorder, or moderate or severe substance or alcohol use disorder [excluding nicotine]).
* Considered to be at significant risk of suicide in the judgment of the Investigator. This includes participants who are actively suicidal (eg, any suicide attempts during the parent study) or are at serious suicidal risk as indicated by any current suicidal intent, including a plan, as assessed by the C-SSRS ("Since Last Visit" version, score of "YES" on suicidal ideation Item 4 or 5) and/or based on clinical evaluation by the Investigator; or are homicidal, in the opinion of the Investigator.
* Non-adherent with study medication (took ≤70% of study drug over any 2-week visit interval) or procedures during the parent study.
* Experienced treatment emergent adverse events (TEAEs) considered related to the study medication from the parent study and judged by the Investigator to be clinically significant to render the participant ineligible for enrollment.
* Have an abnormality on ocular examination that would prohibit continued study participation as determined by the Investigator.
* Use of disallowed concomitant medication or therapy that would have been exclusionary in the parent study, may compromise the safety of the participant, and/or confound the interpretation of protocol assessments.
* Considered by the Investigator to be inappropriate for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability assessments based on Treatment Emergent Adverse Events (TEAEs) and validated clinical scales | Up to 54 Weeks
  An AE is any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of trial intervention, whether or not considered related to the trial intervention. Any AE occurring following the start of treatment or occurring before treatment but increasing in severity afterward were counted as treatment-emergent AE (TEAE). Clinically significant abnormalities in Clinical Laboratory Evaluations, ECGs, Vital Signs, Physical and Ophthalmological examinations, Corneal Specular Microscopy, Columbia Suicide Severity Rating Scale (C-SSRS), and Sexual Functioning Questionnaire-14 (CSFQ-14) will be reported as TEAEs.

SECONDARY OUTCOMES:
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total score over time. | Baseline and up to Week 54
  Change from baseline in MADRS total score over time will be reported. The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change from Baseline in the Snaith-Hamilton Pleasure Scale (SHAPS) total score over time | Baseline and up to Week 54
  The SHAPS is a 14-item participant-reported instrument which measures anhedonia. It has been shown to be valid and reliable in normal and clinical samples, with adequate construct validity, satisfactory test-retest reliability, and high internal consistency. The scale will be completed by the participant and reviewed by site personnel qualified to oversee completeness. Each of the 14 items has a set of 4 responses, 2 of which endorse agreement (Definitely Agree, Agree) and 2 of which endorse disagreement (Disagree, Strongly Disagree). A total score can be derived by summing the responses; items answered with strongly agree are coded as 1 while a strongly disagree response will be coded as 4. Therefore, scores on the SHAPS can range from 14 to 56, with higher scores corresponding to higher levels of anhedonia.
Change from Baseline in the Patient Health Questionnaire-9 (PHQ-9) total score over time. | Baseline and up to Week 54
  Change from baseline in PHQ-9 total score over time will be reported. The 9-item PHQ-9 scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) diagnostic criteria for recurrent or single episode major depressive disorder (MDD) criteria and used both as a screening tool and a measure of response to treatment for depression. Each item is rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Change from Baseline in PHQ-9 Anhedonia Item #1 over time. | Baseline and up to Week 54
  The PHQ-9 is a participant-rated assessment scale for the evaluation of depression symptoms over the past 2 weeks. The PHQ-9 is a reliable and valid measure of depression and depression severity. The questionnaire consists of 9 items and each item is scored from 0 to 3. Participants will be asked how often they have been bothered by symptoms over the past 2 weeks (Not at all [0], Several days [1], More than half the time [2], or Nearly every day [3]). Higher scores indicate higher levels of depression.
Change from Baseline in the Hamilton Anxiety Rating Scale (HAM-A) total score over time. | Baseline and up to Week 54
  The HAM-A is a clinician-rated instrument administered to assess severity of anxiety, its improvement during the course of treatment, and the timing of such improvement. This instrument will be completed by qualified and trained Investigator site raters based on a semi-structured interview for his/her assessment of the participant. The scale consists of 14 items. Each item is rated on a scale of 0 (feeling not present) to 4 (very severe prevalence of the feeling). The HAM-A total score is the sum of the 14 items and the score ranges from 0 to 56.
Change from Baseline in the Clinical Global Impression Scale of Severity (CGI-S) | Baseline and up to Week 54
  Change from baseline in the CGI-S total score over time will be reported. The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants. The CGI-S permits a global evaluation of the participant's condition at a given time.
Clinical Global Impression Scale of Improvement (CGI-I) score at each timepoint | Baseline and up to Week 54
  The CGI-I scale is a clinician-rated instrument that measures the improvement of the participant's symptoms of depression. It is a 7-point scale where a score of 1 indicates that the participant is "very much improved," a score of 4 indicates that the participant has experienced "no change," and a score of 7 indicates that the participant is "very much worse."
Percentage of participants whose MADRS total score decreased by greater than or equal to 50% from Baseline over time | Up to Week 54
Percentage of participants whose MADRS total score decreased to 10 or less over time | Up to Week 54
Change from baseline in the Sheehan Disability Scale (SDS) over time | Baseline and up to Week 54
  The SDS is a participant-rated instrument which was developed to assess functional impairment in 3 related domains of work/school, social, and family life. It is a brief self rated tool where the participant rates the 3 items on an anchored 10 point visual analog scale. Following the participant's self assessment, the rater should review the Work/School and Days Lost items to confirm appropriateness of the selected rating by evaluating the impact of MDD symptoms across those sectors. The SDS may be administered via telephone assessment; however, the participant must be provided with a portable document format (PDF) copy of the assessment for reference of the visual analog scale when selecting their ratings.

CONTACTS AND LOCATIONS:
Locations (153):
- United States (109):
  - Neumora Investigator site, Huntsville, Alabama
  - Neumora Investigator Site, Phoenix, Arizona
  - Neumora Investigator Site, Bentonville, Arkansas
  - Neumora Investigator Site #1, Little Rock, Arkansas
  - Neumora Investigator site, Little Rock, Arkansas
  - Neumora Investigator Site, Rogers, Arkansas
  - Neumora Investigator site, Bellflower, California
  - Neumora Investigator Site, Cerritos, California
  - Neumora Investigator Site, Encino, California
  - Neumora Investigator Site, Garden Grove, California
  - Neumora Investigator Site, Glendale, California
  - Neumora Investigator Site, Imperial, California
  - Neumora Investigator Site, Irvine, California
  - Neumora Investigator Site, Lafayette, California
  - Neumora Investigator Site #1, Long Beach, California
  - Neumora Investigator site, Long Beach, California
  - Neumora Investigator Site, Los Angeles, California
  - Neumora Investigator Site, Newport Beach, California
  - Neumora Investigator Site, Oceanside, California
  - Neumora Investigator Site #1, Orange, California
  - Neumora Investigator Site, Orange, California
  - Neumora Investigator Site, Riverside, California
  - Neumora Investigator Site, San Diego, California
  - Neumora Investigator Site, San Francisco, California
  - Neumora Investigator Site, San Jose, California
  - Neumora Investigator Site, Santa Ana, California
  - Neumora Investigator Site, Sherman Oaks, California
  - Neumora Investigator Site, Temecula, California
  - Neumora Investigator Site, Torrance, California
  - Neumora Investigator Site, Colorado Springs, Colorado
  - Neumora Investigator Site, New Haven, Connecticut
  - Neumora Investigator Site, Norwalk, Connecticut
  - Neumora Investigator Site, Bradenton, Florida
  - Neumora Investigator Site, Brandon, Florida
  - Neumora Investigator Site, Gainesville, Florida
  - Neumora Investigator Site, Hallandale, Florida
  - Neumora Investigator Site, Hialeah, Florida
  - Neumora Investigator Site, Hollywood, Florida
  - Neumora Investigator Site, Jacksonville, Florida
  - Neumora Investigator Site, Lauderhill, Florida
  - Neumora Investigator Site, Maitland, Florida
  - Neumora Investigator Site, Miami, Florida
  - Neumora Investigator site, Miami, Florida
  - Neumora Investigator Site, Miami Beach, Florida
  - Neumora Investigator site, Miami Lakes, Florida
  - Neumora Investigator Site #1, Miami Lakes, Florida
  - Neumora Investigator Site #2, Miami Lakes, Florida
  - Neumora Investigator Site, Miami Springs, Florida
  - Neumora Investigator Site #1, Orlando, Florida
  - Neumora Investigator site, Orlando, Florida
  - Neumora Investigator Site, Orlando, Florida
  - Neumora Investigator Site, Pembroke Pines, Florida
  - Neumora Investigator Site #1, Pompano Beach, Florida
  - Neumora Investigator Site, Pompano Beach, Florida
  - Neumora Investigator Site, Saint Augustine, Florida
  - Neumora Investigator Site, Tampa, Florida
  - Neumora Investigator Site #1, Tampa, Florida
  - Neumora Investigator Site, Atlanta, Georgia
  - Neumora Investigator Site #1, Atlanta, Georgia
  - Neumora Investigator Site, Decatur, Georgia
  - Neumora Investigator Site, Marietta, Georgia
  - Neumora Investigator Site, Savannah, Georgia
  - Neumora Investigator Site, Chicago, Illinois
  - Neumora Investigator Site, Warrenville, Illinois
  - Neumora Investigator Site, Marrero, Louisiana
  - Neumora Investigator Site, New Orleans, Louisiana
  - Neumora Investigator Site, Baltimore, Maryland
  - Neumora Investigator site, Towson, Maryland
  - Neumora Investigator Site, Boston, Massachusetts
  - Neumora Investigator site, Methuen, Massachusetts
  - Neumora Investigator site, Springfield, Massachusetts
  - Neumora Investigator Site, Watertown, Massachusetts
  - Neumora Investigator site, Bloomfield Township, Michigan
  - Neumora Investigator Site, Mankato, Minnesota
  - Neumora Investigator Site, Flowood, Mississippi
  - Neumora Investigator Site, Saint Charles, Missouri
  - Neumora Investigator Site, St Louis, Missouri
  - Neumora Investigator Site, Las Vegas, Nevada
  - Neumora Investigator Site, Berlin, New Jersey
  - Neumora Investigator site, Princeton, New Jersey
  - Neumora Investigator Site, Toms River, New Jersey
  - Neumora Investigator Site, Albuquerque, New Mexico
  - Neumora Investigator Site, Brooklyn, New York
  - Neumora Investigator Site, Buffalo, New York
  - Neumora Investigator Site, Cedarhurst, New York
  - Neumora Investigator Site, Inwood, New York
  - Neumora Investigator Site, New York, New York
  - Neumora Investigator Site, Staten Island, New York
  - Neumora Investigator Site, The Bronx, New York
  - Neumora Investigator Site, Charlotte, North Carolina
  - Neumora Investigator Site, Monroe, North Carolina
  - Neumora Investigator Site, Columbus, Ohio
  - Neumora Investigator Site, Dayton, Ohio
  - Neumora Investigator Site, North Canton, Ohio
  - Neumora Investigator Site, Edmond, Oklahoma
  - Neumora Investigator Site, Oklahoma City, Oklahoma
  - Neumora Investigator Site, Allentown, Pennsylvania
  - Neumora Investigator Site, Media, Pennsylvania
  - Neumora Investigator Site, Philadelphia, Pennsylvania
  - Neumora Investigator Site, Memphis, Tennessee
  - Neumora Investigator Site, Austin, Texas
  - Neumora Investigator site, Austin, Texas
  - Neumora Investigator Site, Dallas, Texas
  - Neumora Investigator Site, Fort Worth, Texas
  - Neumora Investigator Site #1, Houston, Texas
  - Neumora Investigator Site, Houston, Texas
  - Neumora Investigator Site, Wichita Falls, Texas
  - Neumora Investigator Site, Bellevue, Washington
  - Neumora Investigator Site #1, Everett, Washington
- Brazil (7):
  - Neumora Investigator Site, Curitiba, Paraná
  - Neumora Investigator Site, Botafogo - Rio de Janeiro, Rio de Janeiro
  - Neumora Investigator Site, Porto Alegre, Rio Grande do Sul
  - Neumora Investigator Site, Santa Cecília, São Paulo
  - Neumora Investigator Site, São Bernardo do Campo, São Paulo
  - Neumora Investigator Site, São José do Rio Preto, São Paulo
  - Neumora Investigator Site, São Paulo
- Bulgaria (6):
  - Neumora Investigator Site, Cherven Bryag, Pleven
  - Neumora Investigator Site, Sofia, Sofia-Grad
  - Neumora Investigator Site, Varosha, Targovishte
  - Neumora Investigator Site, Kardzhali
  - Neumora Investigator Site, Pleven
  - Neumora Investigator Site, Varna
- Canada (5):
  - Neumora Investigator Site, Kelowna, British Columbia
  - Neumora Investigator Site, Hamilton, Ontario
  - Neumora Investigator Site, Markham, Ontario
  - Neumora Investigator Site, Mississauga, Ontario
  - Neumora Investigator Site, Toronto, Ontario
- Chile (2):
  - Neumora Investigator Site, Santiago, Santiago Metropolitan
  - Neumora Investigator Site, Antofagasta
- Czechia (5):
  - Neumora Investigator Site, Pilsen, Plzeň
  - Neumora Investigator Site, Prague, Prague
  - Neumora Investigator Site, Kladno, South Bohemian
  - Neumora Investigator Site, Kladno
  - Neumora Investigator Site, Prague
- Finland (3):
  - Neumora Investigator Site, Helsinki, Etelä-Suomen Lääni
  - Neumora Investigator Site, Turku, Etelä-Suomen Lääni
  - Neumora Investigator Site, Oulu, Oulun Lääni
- France (5):
  - Neumora Investigator Site, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Neumora Investigator Site, Douai, Hauts-de-France
  - Neumora Investigator Site, Montpellier, Hérault
  - Neumora Investigator Site, La Roche-sur-Yon, Vendée
  - Neumora Investigator Site, Poitiers, Vienne
- Germany (3):
  - Neumora Investigator Site #1, Berlin
  - Neumora Investigator Site, Berlin
  - Neumora Investigator Site, Hamburg
- Poland (6):
  - Neumora Investigator Site, Suchy Las, Greater Poland Voivodeship
  - Neumora Investigator Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Neumora Investigator Site, Wroclaw, Lower Silesian Voivodeship
  - Neumora Investigator Site, Lublin, Lublin Voivodeship
  - Neumora Investigator Site, Białystok, Podkarpackie Voivodeship
  - Neumora Investigator Site, Gdansk, Pomeranian Voivodeship
- Sweden (2):
  - Neumora Investigator Site, Lund, Skåne County
  - Neumora Investigator Site, Stockholm, Stolkholm Ian

IPD SHARING:
Plan to Share IPD: No